CLINICAL TRIAL: NCT02838420
Title: Randomized, Multicenter, Phase III, Open-Label Study of Alectinib Versus Crizotinib in Asian Patients With Treatment-Naive Anaplastic Lymphoma Kinase-Positive Advanced Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate and Compare the Efficacy and Safety of Alectinib Versus Crizotinib and to Evaluate the Pharmacokinetics of Alectinib in Asian Participants With Treatment-Naive Anaplastic Lymphoma Kinase (ALK)-Positive Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO29449
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Anaplastic Lymphoma Kinase-positive Non-small Cell Lung Cancer
MeSH Terms: interventions — alectinib; Crizotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alectinib (Experimental): Participants will receive alectinib capsules orally at a dose of 600 mg BID with food until disease progression, unacceptable toxicity withdrawal of consent, or death.
  Interventions: Drug: Alectinib
- Crizotinib (Active Comparator): Participants will receive crizotinib capsules orally at a dose of 250 mg BID with or without food until disease progression, unacceptable toxicity withdrawal of consent, or death.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Alectinib — Alectinib capsules will be administered orally at a dose of 600 mg BID until disease progression, unacceptable toxicity withdrawal of consent, or death.
  Other Names: RO5424802
  Arms: Alectinib
Drug: Crizotinib — Crizotinib capsules will be administered orally at a dose of 250 mg BID until disease progression, unacceptable toxicity withdrawal of consent, or death.
  Arms: Crizotinib

SUMMARY:
This randomized, multicenter, Phase III, open-label study will evaluate the efficacy and safety of alectinib versus crizotinib and to evaluate the pharmacokinetics of alectinib in asian participants with treatment-naive ALK-positive advanced NSCLC. Participants will be randomized 2:1 into one of the two treatment groups to receive either alectinib (600 milligrams [mg] twice daily [BID]) or crizotinib (250 mg BID) orally, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC that is ALK-positive as assessed by the Ventana immunohistochemistry (IHC) test. Sufficient tumor tissue available to perform ALK IHC is required. Ventana IHC testing will be performed at the designated central laboratory
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
* No history of receiving systemic treatment for advanced, recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC
* Adequate hematologic function: Platelet count greater than equal to (>=) 100×10^9 per liter (/L); absolute neutrophil count (ANC) >=1500 cells per microliter (cells/mcL); hemoglobin>=9.0 grams per deciliter (g/dL)
* Adequate renal function: an estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) formula of >=45 milliliters per minute per 1.73 square meter
* Participants must have recovered from effects of any major surgery or significant traumatic injury at least 28 days before receiving the first dose of study treatment
* Measurable disease (by Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) before administration of study treatment
* Previous brain or leptomeningeal metastases are allowed if the participant is asymptomatic (e.g., diagnosed incidentally at study baseline). Asymptomatic central nervous system (CNS) lesions may be treated at the discretion of the investigator as per local clinical practice. If participant has neurological symptoms or signs because of CNS metastasis, the participant must complete whole-brain radiation or gamma knife irradiation treatment. In all cases, radiation treatment must be completed >=14 days before enrollment and disease must be clinically stable
* For all females of childbearing potential, a negative serum pregnancy test result must be obtained within 3 days prior to starting study treatment
* For women who are not postmenopausal (>=12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus), agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 3 months after the last dose of study drug. Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Examples of contraceptive methods with a failure rate of <1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide
* For men, agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 3 months after the last dose of study drug. Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* A malignancy within the previous 3 years (other than curatively treated basal cell carcinoma of the skin, early gastrointestinal (GI) cancer by endoscopic resection, in situ carcinoma of the cervix, or any cured cancer that is considered to have no impact in progression-free survival (PFS) or overall survival (OS) for the current NSCLC)
* Any GI disorder that may affect absorption of oral medications, such as malabsorption syndrome or status post-major bowel resection
* Liver disease characterized by:
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than (>) 3× the upper limit of normal (ULN; >=5×ULN for participants with concurrent liver metastases) confirmed on two consecutive measurements; or
* Impaired excretory function (e.g., hyperbilirubinemia), synthetic function, or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices; or
* Acute viral or active autoimmune, alcoholic, or other types of hepatitis
* National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 Grade 3 or higher toxicities because of any previous therapy (e.g., radiotherapy) (excluding alopecia), which have not shown improvement and are strictly considered to interfere with current study medication
* History of organ transplant
* Co-administration of anti-cancer therapies other than those administered in this study
* Baseline QTc >470 ms or symptomatic bradycardia
* Administration of strong/potent cytochrome P4503A inhibitors or inducers within 14 days prior to the receiving the first dose of study treatment and during treatment with alectinib or crizotinib
* Administration of agents with potential QT interval prolonging effects within 14 days prior to receiving the first dose of study drug
* History of hypersensitivity to any of the additives in the alectinib or crizotinib drug formulation
* Pregnant or lactating
* Known human immunodeficiency virus (HIV-positivity or acquired immunodeficiency syndrome (AIDS)-related illness
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or the absorption of oral medications or that would, in the opinion of the Principal Investigator, pose an unacceptable risk to the participant in this study
* Any psychological, familial, sociological, or geographical condition that potentially hampers compliance with the study protocol requirements or follow-up procedures; those conditions should be discussed with the participant before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- China (15):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai chest hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
- South Korea (3):
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Thailand (3):
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Zhou C, Kim SW, Reungwetwattana T, Zhou J, Zhang Y, He J, Yang JJ, Cheng Y, Lee SH, Bu L, Xu T, Yang L, Wang C, Liu T, Morcos PN, Lu Y, Zhang L. Alectinib versus crizotinib in untreated Asian patients with anaplastic lymphoma kinase-positive non-small-cell lung cancer (ALESIA): a randomised phase 3 study. Lancet Respir Med. 2019 May;7(5):437-446. doi: 10.1016/S2213-2600(19)30053-0. Epub 2019 Apr 10. PMID 30981696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Asian adult participants with treatment-naive anaplastic lymphoma kinase (ALK)-positive advanced, recurrent, or metastatic non-small cell lung cancer (NSCLC) were enrolled at 21 study sites in 3 countries - China, Korea, and Thailand.
Groups:
- Alectinib: Participants received alectinib capsules orally at a dose of 600 mg twice a day (BID) with food until disease progression, unacceptable toxicity withdrawal of consent, or death.
- Crizotinib: Participants received crizotinib capsules orally at a dose of 250 mg BID with or without food until disease progression, unacceptable toxicity, withdrawal of consent, or death.
Period: Overall Study
Arm/Group | Alectinib | Crizotinib
Started | 125 | 62
Completed | 0 | 0
Not Completed | 125 | 62
Not completed — Ongoing in Study | 113 | 45
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Death | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alectinib | Crizotinib | Total
Number analyzed (Participants) | 125 | 62 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (11.3) | 51.1 (12.6) | 50.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 28 | 89
  Male | 64 | 34 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 124 | 60 | 184
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 125 | 62 | 187
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Determined by Investigator Using Response Evaluation Criteria in Solid Tumor (RECIST) v1.1
Description: PFS was defined as the time (in months) from randomization to the first documentation of disease progression, as determined by the investigators, or to death from any cause, whichever occurred first.
Time Frame: From the date of randomization to the date of the first documented disease progression or death, whichever occurred first (up to overall period of approximately 40 months)
Population: The primary analysis population for efficacy was the intent-to-treat (ITT) population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 125 | 62
Months | NA [20.3 to NA] — Median and upper bound of 95% CI could not be estimated as PFS had not been reached at the time of data cutoff for the primary end point. | 11.1 [9.1 to 13.0]

2. Secondary Outcome: PFS as Determined by Independent Review Committee (IRC) Using RECIST v1.1
Description: PFS was defined as the time (in months) from randomization to the first documentation of disease progression, as determined by an independent review committee, or to death from any cause, whichever occurred first.
Time Frame: Baseline, Week 8, thereafter every 8 weeks until disease progression, death or withdrawal from the study and 4 weeks after permanent discontinuation (up to overall period of approximately 40 months)
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Participants With Objective Response of Complete Response (CR) or Partial Response (PR) as Determined by Investigator Using RECIST v1.1
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Time to Progression of Disease in the CNS as Determined by IRC Using RECIST v1.1
Time Frame: as for outcome 2
Reporting Status: Not Posted

5. Secondary Outcome: Time to Progression of Disease in the CNS as Determined by IRC Using Response Assessment in Neuro-Oncology (RANO)
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Secondary Outcome: Duration of Response (DOR) Assessed by Investigator Using RECIST v1.1
Time Frame: as for outcome 2
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival Time
Time Frame: Baseline, until death (up to overall period of approximately 40 months)
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Participants With Non-serious Adverse Events and Serious Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to overall period of approximately 40 months
Population: The safety population was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 125 | 62
Percentage of Participants
  Serious Adverse Events | 15.2 | 25.8
  Non-Serious Adverse Events | 99.2 | 100.0

9. Secondary Outcome: Time to Deterioration Assessed Using EORTC Quality of Life Questionnaire-Core (QLQ-C30) Score
Time Frame: Baseline, Week 4, thereafter every 4 weeks until disease progression, death or withdrawal from the study and 4 weeks after permanent discontinuation (up to overall period of approximately 40 months)
Reporting Status: Not Posted

10. Secondary Outcome: Time to Deterioration Assessed Using EORTC Quality of Life Questionnaire-Lung Cancer Module (QLQ-LC13) Score
Time Frame: as for outcome 9
Reporting Status: Not Posted

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of Alectinib and Its Metabolite
Description: AUC was collected for both alectinib and its major metabolite, M4, and was based on their concentrations in plasma over time.
Time Frame: Baseline and Week 4 predose (within 2 hours before administration of study drug)
Population: The PK evaluable population for this outcome measure was a subset of frequent-sampling Chinese participants who received any dose of alectinib, and who had at least one quantifiable post-baseline PK sample available. This outcome measure was specific to the alectinib arm, and no data was collected from participants in the crizotinib arm.
Measure: Mean (Standard Deviation); unit: Hours*nanogram/milliliter (hr*ng/mL)
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 20 | 0
Hours*nanogram/milliliter (hr*ng/mL)
  Alectinib Baseline | 1590 (852) |
  M4 Baseline | 471 (243) |
  Alectinib Week 4 | 7760 (3270) |
  M4 Week 4 | 2890 (1130) |

12. Secondary Outcome: Maximum Plasma Concentration Observed (Cmax) of Alectinib and Its Metabolite
Description: Cmax was collected for both alectinib and its major metabolite, M4, and was based on their concentrations in plasma over time.
Time Frame: Baseline and Week 4 predose (within 2 hours before administration of study drug)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Nanograms/milliliter (ng/mL)
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 20 | 0
Nanograms/milliliter (ng/mL)
  Alectinib Baseline | 255 (130) |
  M4 Baseline | 71.4 (33.5) |
  Alectinib Week 4 | 861 (332) |
  M4 Week 4 | 306 (111) |

13. Secondary Outcome: Time to Cmax (Tmax) of Alectinib and Its Metabolite
Description: Tmax was collected for both alectinib and its major metabolite, M4, and was based on their concentrations in plasma over time.
Time Frame: Baseline and Week 4 predose (within 2 hours before administration of study drug)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour (hr)
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 20 | 0
Hour (hr)
  Alectinib Baseline | 5.61 (3.02) |
  M4 Baseline | 8.19 (2.30) |
  Alectinib Week 4 | 4.30 (2.45) |
  M4 Week 4 | 4.11 (3.06) |

ADVERSE EVENTS:
Time Frame: Up to approximately 40 months
Description: The safety population was defined as all participants who received at least one dose of study drug. All participants in the ITT population received at least one dose of study drug and were included in the safety population.
Arm/Group | Alectinib | Crizotinib
All-Cause Mortality (participants affected / at risk) | 8/125 | 13/62
Serious Adverse Events (participants affected / at risk) | 19/125 | 16/62
Other Adverse Events (participants affected / at risk) | 124/125 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib (N=125) | Crizotinib (N=62)
Lung infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Blood uric acid increased (Investigations) | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Brain ooedema (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Post procedural ooedema (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib (N=125) | Crizotinib (N=62)
Aspartate aminotransferase increased (Investigations) | 65 | 31
Alanine aminotransferase increased (Investigations) | 52 | 34
Blood creatine phosphokinase increased (Investigations) | 55 | 18
Blood bilirubin increased (Investigations) | 61 | 2
Blood alkaline phosphatase increased (Investigations) | 33 | 8
Blood creatinine increased (Investigations) | 25 | 15
Bilirubin conjugated increased (Investigations) | 33 | 2
Weight increased (Investigations) | 23 | 2
Gamma-glutamyltransferase increased (Investigations) | 5 | 17
Haemoglobin decreased (Investigations) | 18 | 3
White blood cell count decreased (Investigations) | 6 | 15
Blood lactate dehydrogenase increased (Investigations) | 11 | 7
Neutrophil count decreased (Investigations) | 4 | 12
Blood bilirubin unconjugated increased (Investigations) | 14 | 0
Blood thyroid stimulating hormone increased (Investigations) | 12 | 1
Electrocardiogram QT prolonged (Investigations) | 4 | 7
Blood albumin decreased (Investigations) | 4 | 5
Blood creatine phosphokinase MB increased (Investigations) | 4 | 5
Weight decreased (Investigations) | 1 | 5
Protein total decreased (Investigations) | 0 | 4
Constipation (Gastrointestinal disorders) | 45 | 31
Diarrhoea (Gastrointestinal disorders) | 16 | 31
Nausea (Gastrointestinal disorders) | 8 | 21
Vomiting (Gastrointestinal disorders) | 7 | 22
Fatigue (General disorders) | 11 | 9
Pyrexia (General disorders) | 11 | 9
Chest pain (General disorders) | 10 | 8
Oedema peripheral (General disorders) | 8 | 10
Chest discomfort (General disorders) | 10 | 3
Asthenia (General disorders) | 6 | 5
Oedema (General disorders) | 9 | 2
Sinus bradycardia (Cardiac disorders) | 37 | 11
Bradycardia (Cardiac disorders) | 12 | 5
Upper respiratory tract infection (Infections and infestations) | 23 | 6
Nasopharyngitis (Infections and infestations) | 15 | 3
Urinary tract infection (Infections and infestations) | 8 | 1
Lung infection (Infections and infestations) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 38 | 14
Neutropenia (Blood and lymphatic system disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Decreased appetite (Metabolism and nutrition disorders) | 6 | 22
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 9
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 2
Rash (Skin and subcutaneous tissue disorders) | 21 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 12 | 5
Dizziness (Nervous system disorders) | 7 | 13
Headache (Nervous system disorders) | 7 | 10
Dysgeusia (Nervous system disorders) | 1 | 10
Liver injury (Hepatobiliary disorders) | 14 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 9 | 4
Insomnia (Psychiatric disorders) | 7 | 6
Vision blurred (Eye disorders) | 2 | 9
Haematuria (Renal and urinary disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT02838420/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT02838420/SAP_001.pdf